CLINICAL TRIAL: NCT03118245
Title: A Randomized Comparison of Ambu AuraGain (Original Name of Product) Laryngeal Mask Airway and I-gel in Children
Brief Title: Ambu AuraGain Laryngeal Mask Airway and I-gel in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H1704-083-846
Record Dates: First submitted 2017-04-09; First posted 2017-04-18 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AuraGain group (Experimental): AuraGain is inserted for maintenance of general anesthesia. The size 1 is for children <5kg, size 2 for 5-10kg, size 2 for 10-20kg, and size 2.5 for 20-30kg.
  Interventions: Device: AuraGain
- I-gel group (Experimental): I-gel is s inserted for maintenance of general anesthesia. The size 1 is for children weighted 2-5kg, size 2 for 5-12kg, size 2 for 10-25kg, and size 2.5 for 25-35kg.
  Interventions: Device: I-gel

INTERVENTIONS:
Device: AuraGain — After anesthetic induction, AuraGain is inserted in children
  Other Names: Ambu AuraGain
  Arms: AuraGain group
Device: I-gel — After anesthetic induction, I-gel is inserted in children
  Other Names: I-gel supraglottic airway
  Arms: I-gel group

SUMMARY:
Children aged below 7 years are randomly assigned to AuraGain Group or I-gel group. After anesthetic induction, AuraGain or I-gel is inserted and mechanical ventilation is started. Oropharyngeal leak pressure, peak inspiratory pressure, success rate for insertion, ease for insertion, ease for gastric tube insertion and fiberoptic bronchoscopic views will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children < 7 years old who scheduled for general anesthesia using supraglottic airway

Exclusion Criteria:

* Children who require tracheal intubation
* Emergency operation without nil per os
* History of C-spine surgery or disease
* History of Esophageal disease or surgery

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 30 seconds after AuraGain or I-gel insertion
  The airway pressure at which a leak sound is detected around the patient's mouth and at which the airway pressure has reached equilibrium, when the pressure-limiting valve of the anesthesia breathing system is closed and the fresh gas flow rate is fixed at 3 liter/min

SECONDARY OUTCOMES:
Peak inspiratory pressure | through study completion, an average of 1 hour
  Peak airway pressure
Success rate | Within 5 minutes after anesthetic induction
  Success rate of AuraGain or I-gel insertion
Ease of AuraGain or I-gel insertion | Within 5 minutes after anesthetic induction
  1. No resistance 2. Moderate resistance 3. High resistance 4. Inability to pass
Ease of gastric tube insertion | Within 5 minutes after anesthetic induction
  1. Easy 2. Difficult 3. Unable to pass
fiberoptic bronchoscopic veiw | Within 10 minutes after anesthetic induction
  1. No visible glottis 2. Visible glottis and anterior epiglottis 3. Visible glottis and posterior epiglottis 4. Only glottis is visible

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided